CLINICAL TRIAL: NCT04143633
Title: Low FODMAP Diet Chronic Effect on Nutritional Status, Disease Activity and Gut Microbiota in Patients With IBS and UC
Brief Title: Low FODMAP Diet on Nutritional Status, Disease Activity and Gut Microbiota in IBS and UC With Normal or Overweight BMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, Nallely Bueno Hernández, Investigator In Medical Science B, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DI/17/301/03/084
Record Dates: First submitted 2019-10-08; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-03

CONDITIONS: IBD - Inflammatory Bowel Disease; IBS - Irritable Bowel Syndrome; UC - Ulcerative Colitis
Keywords: Irritable Bowel Syndrome; Ulcerative Colitis; Low FODMAP diet; Nutritional status; Standard diet
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Colitis, Ulcerative | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient doesn´t know the type of diet (standard or low FODMAP)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FODMAP diet in Irritable Bowel Syndrome (Experimental): Patients with IBS will be randomized to standard diet or low fodmap diet. The nutritional status (body composition and clinical parameters), gut microbiota, adherence to treatment, improvement of gastrointestinal symptoms and quality of life will be evaluated for 10 weeks.
  Interventions: Other: Low FODMAP diet; Other: Standard diet
- FODMAP diet in Ulcerative Colitis (Experimental): Patients with UC will be randomized to standard diet or low fodmap diet. The nutritional status (body composition and clinical parameters), gut microbiota, adherence to treatment, improvement of gastrointestinal symptoms and quality of life will be evaluated for 10 weeks.
  Interventions: Other: Low FODMAP diet; Other: Standard diet
- FODMAP diet in healthy patients (Active Comparator): Healthy patients will be randomized to standard diet or low fodmap diet. The nutritional status (body composition and clinical parameters), gut microbiota, adherence to treatment, improvement of gastrointestinal symptoms and quality of life will be evaluated for 10 weeks.
  Interventions: Other: Low FODMAP diet; Other: Standard diet

INTERVENTIONS:
Other: Low FODMAP diet — The diet will be in accordance to the baseline energy expenditure calculated by Harris-Benedict whit 55% of carbohydrates, 25% of lipids and 20% of proteins, divided in five meals. The distribution of carbohydrates depends on the content of fodmaps on each food.
Other: Standard diet — The diet will be in accordance to the baseline energy expenditure calculated by Harris-Benedict whit 55% of carbohydrates, 25% of lipids and 20% of proteins, divided in five meals. Cruciferous vegetables, fruits and condiments will be eliminated and a normal content of fodmap.

SUMMARY:
Gastrointestinal disorders represents 20-50% of referrals to the gastroenterologist; being the most affected womens, youths and older adults. Among these alterations are the Irritable Bowel Syndrome (IBS) and Ulcerative Colitis (UC), which affects the gut causing impaired motility. The pharmacological and nutritional treatment are modified according to the symptomatology and activity of each patients. Currently the implementation of low FODMAP diets for 6 to 8 weeks in patients whith IBS improves symptoms such as bloating, flatulence and abdominal pain. However due to the number of restricted foods a long term attachment could limited the nutritional content, consequently affecting the nutritional status, gut microbiota an quality of life. A low FODMAP diet are useful to improve gastrointestinal symptoms in patients with UC and causes changes in nutritional status.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) and Ulcerative Colitis (UC) affect principally the gut, causing symptoms that alter intestinal motility, with a multifactorial etiology. The pharmacological and nutritional treatment varies according to the symptoms and activity of each patient. The most commonly used are the standard diet (SD), which excludes foods known as irritants or inflammatory. On the other hand, are the low fodmap diet (LFD) (fermentable oligosaccharides. disaccharides, monosaccharides and polyols), these highly fermentable carbohydrates can pass unabsorbed to the colon and induce the gas production due to the fermentation of gut microbiota and cause symptoms such as: bloating, flatulence, abdominal pain and altered bowel habit. It consists in two stages: first the restriction of all foods that contain fodmaps and second the re exposure in which indicate the introduction of each food restricted before to evaluate the tolerance, for 6 to 8 weeks. Some studies show that the low fodmap diet improve the symptoms in both groups, however because of the restriction and the limited content of foods, they have had risk to present nutritional deficiencies. The aim of the present is to evaluate the effect of a low fodmap diet for 10 weeks on gastrointestinal symptoms, nutritional status and microbiota in patients with IBS and UC.

Methods: a controlled, blinded clinical trial will be conducted in patients who assist to medical monitoring in gastroenterology service with diagnosis of IBS or UC. The sample size was determined with a 0.5 effect size, an alpha error 0.05 and power of 80%, which determined 64 patients for each group (total: 128). After singing the informed consent, will be determined their total energy expenditure (TEE) and consecutively will be assigned an ID previously randomized to SD (<16 g of fodmaps) or LFD (<10 g of fodmaps), with a distribution of 55% carbohydrates, 20% proteins and 25% lipids. During the 10 weeks will be three follow-ups, first the basal, intermediate (week 5) and final (10 weeks after), will be performed body composition (RJL Quantum III), anthropometry (waist, hip, arm and chest circumference), gastrointestinal symptoms (ROMA III and Mayo Scale), quality of life (WHOQL-BREF), food frequency and 24-hour reminder and blood chemistry (anemia, hypoalbuminemia, vitamin D, calcium, potassium, c reactive protein, VSG, etc), all of them basal and final.

ELIGIBILITY:
Inclusion Criteria:

* Irritable Bowel Syndrome confirmed by Rome criteria III
* Ulcerative Colitis confirmed by Mayo Scale
* Informed Consent signed
* BMI between 18.5 and 29.9 kg/m2
* Males and females
* Age between 18-59 years
* Mexican patients

Exclusion Criteria:

* Chron´s disease diagnosed
* Treatment whith antibiotis during the last two weeks
* Bowel resection
* Short bowel syndrome
* Treatment wihth probiotics or enzimes (A-galactosidase)
* Pregnancy
* Nutritional deficiencies or anemia
* Patients whith diet supplements

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Nutritional status | The patients will be evaluated at weeks 1 and 10
  Changes from baseline of nutrtitional status measured with cholesterol (mg/dl), triglycerides (mg/dl), albumin (mg/dl), calcium (mg/dl), iron (mg/dl), vitamin B12 (mg/dl), vitamin D (mg/dl), hemoglobin (mg/dl), hematocrit (mg/dl), creatinin (mg/dl) on blood

SECONDARY OUTCOMES:
Quality of life in patients with Irritable Bowel Syndrome and Inflammatory Bowel Disease | The patients will be evaluated at weeks 1, 5 and 10
  Changes from baseline of WHOQOL- BREF (World Health Organization Quality of Life) questionary score (the higher score, the higher quality of life represents) measured with a Likert scale at 10 weeks of nutritional intervention in patients wiht irritable bowel syndrome and inflammatory bowel disease
Adherence to treatment | The patients will be evaluated at weeks 1, 5 and 10
  By 24 hour recalls during the ten weeks of the study and food frequencies at week one, five and ten.
Body composition analysis | The patients will be evaluated at weeks 1, 5 and 10
  Changes from baseline of the percentage of body fat (%), muscle (%) and water (%) at 10 weeks of nutritional intervention, using RJL System IV
Gut microbiota with a low FODMAP diet | Participants will be evaluated at weeks 1, 5 and 10
  The patient will be asked for a stool sample before and after the diet, the microbiota were measure by PCR
Blood chemistry | Participants will be evaluated at weeks 1 and 10
  Changes from baseline glucose, creatinine, high density lipoproteins, low density lipoproteins, cholesterol levels (mg/dL) at 10 weeks of nutritional intervention in patients with IBS and IBD
Irritable Bowel Syndrome Severity Score | Participants will be evaluated at weeks 1, 5 and 10
  Changes from baseline in the presence or absence of gastrointestinal symptoms where the higher the score, more severity of symptoms are assesed using a percentage scale 0-100%, at 10 weeks with low FODMAP diet in patients wih IBS and IBD
Gastrointestinal Symptoms Severity | Participants will be evaluated at weeks 1, 5 and 10
  Changes from baseline of presence or abscense of gastrointestinal symptoms where the higher the score, the higher severity of symptoms (assesed using cualitative scale with options ranging from minimal symptoms to very annoying symptoms) at 10 weeks with low FODMAP diet in patients wih IBS and IBD
Anthropometric measurements | Participants will be evaluated at weeks 1, 5 and 10
  Changes from baseline of arm, waist and hips circumferences in centimeters at 12 weeks of nutritional intervention in patientes with IBS anda IBD

CONTACTS AND LOCATIONS:
Overall Officials: Nallely Bueno Hernádez, PhD, Principal Investigator — Hospital General de México
Locations (1):
- Nallely Bueno Hernández, Mexico City, Cuauhtémoc, Mexico